CLINICAL TRIAL: NCT07110701
Title: A Comparative Clinical Evaluation of Two Resin-Based Fissure Sealants Applied With Different Isolation Techniques: An 18-Month Follow-Up Study
Brief Title: Clinical Evaluation Fissure Sealants Applied With Different Isolation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ebru KUCUKYİLMAZ, Prof. Dr., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025/059
Record Dates: First submitted 2025-07-03; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Fissure Sealant; Rubberdam; Isolation
Keywords: Resin-Based Fissure Sealants; isolation techniques; rubberdam

STUDY DESIGN:
Intervention Model Description: The randomized, controlled, single-blind clinical study
Who Masked: Outcomes Assessor
Masking Description: A split-mouth study design was implemented, in which two distinct fissure sealant materials were applied using two different isolation techniques. Each participant received both types of sealants-one placed under rubber dam isolation and the other under cotton roll isolation. To reduce the risk of allocation bias, the assignment of sealant materials and isolation methods to specific teeth was randomized. A computer-generated randomization list (Research Randomizer, Version 4.0) was used to determine both the order of sealant application and the side (right or left mandibular molar) to which each material would be assigned. Based on the combination of sealant type and isolation method, this process resulted in the creation of four distinct study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- a highly filled fluoride-containing fissure sealant with rubber dam isolation (Active Comparator): Plaque and debris were meticulously removed from the occlusal surfaces using a rotary brush in conjunction with a non-fluoridated prophylactic paste. In accordance with the randomization protocol, and subsequent to the allocation of materials and isolation techniques for each quadrant, individual teeth were isolated using a rubber dam to ensure optimal protection against salivary contamination. All clinical procedures were performed under standardized illumination and strictly adhered to the manufacturers' guidelines. The polymerization of the highly filled, fluoride-releasing fissure sealant was executed using a calibrated LED light-curing unit. Following application, each sealant was rigorously assessed for the absence of air entrapment, quality of marginal adaptation, retention, and the adequacy of polymerization.
  Interventions: Other: Retention of the fissure sealants evaluated
- a highly filled fluoride-containing fissure sealant with cotton roll isolation, (Active Comparator): Plaque and debris were meticulously removed from the occlusal surfaces using a rotary brush in combination with a non-fluoridated prophylactic paste. In line with the randomization protocol and subsequent allocation of the materials and isolation methods for each side of the patient, individual teeth were isolated using cotton rolls in conjunction with high-volume suction to minimize the risk of salivary contamination. All procedures were performed under standardized illumination and strictly followed the manufacturers' instructions. Polymerization of the highly filled, fluoride-releasing fissure sealant was carried out using a calibrated LED light-curing unit. Following application, each sealant was carefully evaluated for the presence of air voids, the quality of marginal adaptation, retention, and the completeness of polymerization.
  Interventions: Other: Retention of the fissure sealants evaluated
- an unfilled fluoride-containing fissure sealant with rubber dam isolation, (Active Comparator): Plaque and debris were meticulously removed from the occlusal surfaces using a rotary brush in conjunction with a non-fluoridated prophylactic paste. In accordance with the randomization protocol and following the allocation of materials and isolation methods for each side of the patient, individual teeth were isolated using a rubber dam to ensure effective prevention of salivary contamination. All clinical procedures were performed under standardized illumination and in strict compliance with the manufacturers' instructions. Polymerization of the unfilled, fluoride-releasing fissure sealant was performed using a calibrated LED light-curing unit. Following the application, each sealant was thoroughly evaluated for the presence of air voids, marginal adaptation, retention, and completeness of polymerization.
  Interventions: Other: Retention of the fissure sealants evaluated
- an unfilled fluoride-containing fissure sealant with cotton roll isolation. (Active Comparator): Plaque and debris were meticulously removed from the occlusal surfaces using a rotary brush in combination with a non-fluoridated prophylactic paste. In line with the randomization protocol and subsequent determination of the materials and isolation techniques for each side of the patient, individual teeth were isolated using cotton rolls in conjunction with high-volume suction to minimize salivary contamination. All procedures were carried out under standardized illumination and in strict accordance with the manufacturers' recommendations. Polymerization of the unfilled, fluoride-releasing fissure sealant was performed using a calibrated LED light-curing unit. Following each application, the sealant was thoroughly evaluated for the presence of air voids, quality of marginal adaptation, retention, and completeness of polymerization.
  Interventions: Other: Retention of the fissure sealants evaluated

INTERVENTIONS:
Other: Retention of the fissure sealants evaluated — Following classification system was employed for the retention evaluation of the sealants: 1 = complete retention; 2 = partial loss; or 3 = complete loss.

SUMMARY:
The aim of this clinical study was to evaluate the effects of different isolation methods and material filler ratios on the retention rates of two different fluoride-containing fissure sealants over an 18-month period.

Methods:

A total of 100 children (200 teeth) participated in this randomized, single-blind, split-mouth clinical trial. The mandibular permanent first molars of each participant were divided into two groups: one receiving a highly filled fluoride-releasing fissure sealant (Fissurit FX, Voco, Germany), and the other an unfilled fluoride-releasing sealant (Teethmate F-1, Kuraray, Germany). Each material group was also divided into two subgroups based on the isolation method used: rubber dam or cotton roll isolation. Sealant retention rates were evaluated at 6-, 12-, and 18-month follow-up visits. Data were statistically analyzed using a 0.05 significance level.

DETAILED DESCRIPTION:
The aim of this randomized, controlled clinical trial was to assess (i) the retention rates of two different resin-based fissure sealant materials-one containing a high filler content and the other unfilled, both fluoride-releasing-and (ii) the effect of the isolation method (rubber dam versus cotton roll isolation) on sealant retention. Additionally, the study evaluated the effectiveness of these materials and isolation techniques in the prevention of dental caries. The null hypotheses tested were: (i) there is no significant difference in the retention rates between the two types of resin-based fissure sealants, and (ii) the type of isolation method employed does not significantly influence sealant retention.

Study Design:

This randomized, controlled, single-blind clinical trial was approved by the Medical Ethics Committee of Izmir Katip Celebi University (Approval No: 2025/059). Prior to the commencement of treatment, written informed consent was obtained from the parents or legal guardians of all participants. The study was conducted in accordance with the CONSORT (Consolidated Standards of Reporting Trials) guidelines to ensure the transparency and integrity of the methodology and results.

The study included 100 healthy children between the ages of 6 and 12 years (mean age: 7.9 years), all classified as ASA Class I (American Society of Anesthesiologists) and exhibiting cooperative behavior, as determined by a Frankl Behavior Rating Scale score of 3 or 4. All participants had fully erupted mandibular first permanent molars on both sides (totaling 200 teeth) requiring the application of pit-and-fissure sealants.

The clinical procedures were conducted by two trained investigators: one responsible for the baseline examination and treatment, and the other-blinded to the materials and methods used-responsible for follow-up assessments. Examiner calibration was performed at 20 randomly selected sites, and agreement was considered acceptable upon achieving substantial inter-examiner reliability (Cohen's Kappa ≥ 0.7).

Prior to enrollment, 178 children were screened by the primary operator, who assessed caries presence using visual inspection based on ICDAS criteria. Participants' medical and dental histories were recorded, and a clinical examination was performed using a blunt explorer and mouth mirror. Radiographic evaluation, including bilateral bitewing radiographs, was conducted to ensure the absence of dental caries in the target molars.

Caries risk assessment was performed using the Cariogram software (CarEng, version 3.0, Malmö University, Sweden). Factors included in the risk profile were: caries experience (DMFT/DMFS indices, new caries within the past year, existing restorations and missing teeth), presence of systemic conditions, dietary habits (particularly sugar intake), frequency of meals and snacks, Silness-Löe Plaque Index scores, Streptococcus mutans levels in saliva (assessed via strip test), fluoride exposure, salivary flow rate (stimulated saliva test), and salivary buffer capacity (measured using Saliva-Check Buffer or equivalent strip tests). Only patients identified as having a moderate risk of caries were included.

Eligible participants were enrolled following informed consent and child assent. Evaluation of the pit-and-fissure sealants was conducted at 6-, 12-, and 18-month recall appointments to monitor the presence of carious lesions and sealant retention. Assessments were performed by a calibrated pediatric dentist who remained blinded to the materials used. Prior to evaluation, teeth were cleaned with a toothbrush, air-dried, and examined under appropriate illumination. Caries lesions were recorded using the ICDAS II criteria, and sealant retention was classified as follows:

1. = Complete retention
2. = Partial loss
3. = Complete loss

Sealants exhibiting complete loss at any recall visit were re-applied; however, such teeth were withdrawn from further statistical analysis and recorded as failures throughout the remainder of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* The study comprised 100 healthy children aged between 6 and 12 years
* ASA class I (American Society of Anesthesiologists),
* exhibit cooperative behavior with a score of 3 or 4 on the Frankl Behavior Rating Scale.
* All participants has to be fully erupted lower first permanent molars on both sides (200 teeth), which required the application of pit and fissure sealants.
* The inclusion criteria is based on the International Caries Detection and Assessment System II (ICDAS II) criteria, including deep and retained pits and fissures, no restorations, and no evidence of caries lesions

Exclusion Criteria:

* Participants with special needs or systemic disease (ASA classification II or higher),
* requiring emergency dental care,
* suffering from a severe gag reflex or an allergy to latex,
* exhibiting uncooperative behavior (Frankl Score 1 or 2),
* exhibiting molars with anomalies of the enamel/dentin, or
* unable to attend follow-up appointments were excluded from the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
The retention rates of two different resin-based fissure sealant materials (a pit and fissure sealant containing high-filler fluoride and a pit and fissure sealant containing non-filler fluoride) | The evaluation of pit-and-fissure sealants was conducted to record the presence of caries lesions and sealant retention at 6-, 12-, and 18-month follow-up visits.
  Following classification system was employed for the retention evaluation of the sealants: 1 = complete retention; 2 = partial loss; or 3 = complete loss.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hicks MJ, Flaitz CM. Epidemiology of dental caries in the pediatric and adolescent population: a review of past and current trends. J Clin Pediatr Dent. 1993 Fall;18(1):43-9. PMID 8110613
- [Background] Brown LJ, Kaste LM, Selwitz RH, Furman LJ. Dental caries and sealant usage in U.S. children, 1988-1991: selected findings from the Third National Health and Nutrition Examination Survey. J Am Dent Assoc. 1996 Mar;127(3):335-43. doi: 10.14219/jada.archive.1996.0203. PMID 8819780
- [Background] Bahrololoomi Z, Soleymani A, Heydari Z. In vitro comparison of microleakage of two materials used as pit and fissure sealants. J Dent Res Dent Clin Dent Prospects. 2011 Summer;5(3):83-6. doi: 10.5681/joddd.2011.019. Epub 2011 Sep 5. PMID 22991611
- [Background] Deery C. Caries detection and diagnosis, sealants and management of the possibly carious fissure. Br Dent J. 2013 Jun;214(11):551-7. doi: 10.1038/sj.bdj.2013.525. PMID 23744208
- [Background] Ripa LW. Sealants revisted: an update of the effectiveness of pit-and-fissure sealants. Caries Res. 1993;27 Suppl 1:77-82. doi: 10.1159/000261608. PMID 8500131
- [Background] Ahovuo-Saloranta A, Hiiri A, Nordblad A, Worthington H, Makela M. Pit and fissure sealants for preventing dental decay in the permanent teeth of children and adolescents. Cochrane Database Syst Rev. 2004;(3):CD001830. doi: 10.1002/14651858.CD001830.pub2. PMID 15266455
- [Background] Feigal RJ. The use of pit and fissure sealants. Pediatr Dent. 2002 Sep-Oct;24(5):415-22. PMID 12412955
- [Background] Beauchamp J, Caufield PW, Crall JJ, Donly K, Feigal R, Gooch B, Ismail A, Kohn W, Siegal M, Simonsen R; American Dental Association Council on Scientific Affairs. Evidence-based clinical recommendations for the use of pit-and-fissure sealants: a report of the American Dental Association Council on Scientific Affairs. J Am Dent Assoc. 2008 Mar;139(3):257-68. doi: 10.14219/jada.archive.2008.0155. PMID 18310730
- [Background] Alhareky MS, Mermelstein D, Finkelman M, Alhumaid J, Loo C. Efficiency and patient satisfaction with the Isolite system versus rubber dam for sealant placement in pediatric patients. Pediatr Dent. 2014 Sep-Oct;36(5):400-4. PMID 25303507

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT07110701/Prot_SAP_ICF_000.pdf